CLINICAL TRIAL: NCT05606393
Title: Establishment of Virtual Reality System for Stroke Patients With Aphasia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-01-012C
Record Dates: First submitted 2022-11-01; First posted 2022-11-04 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Aphasia
Keywords: virtual reality; aphasia; language rehabilitation; stroke
MeSH Terms: conditions — Aphasia; Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- traditional speech therapy and additional virtual reality training group (Experimental): Each participant received 1-hour traditional speech therapy(ST) and additional 30-minute VR training immediately after each session of traditional ST. All participants received 3 sessions of treatment every week for 3 weeks.
  Interventions: Other: virtual reality speech training; Other: traditional speech therapy
- traditional speech therapy group (Active Comparator): Each participant received 1-hour traditional speech therapy(ST) only for each session. All participants received 3 sessions of treatment every week for 3 weeks.
  Interventions: Other: traditional speech therapy

INTERVENTIONS:
Other: virtual reality speech training — virtual reality speech training that focuses on receptive and expressive aspects of language, through a newly developed interactive virtual reality software
  Arms: traditional speech therapy and additional virtual reality training group
Other: traditional speech therapy — traditional speech therapy in current clinical use, that focuses on language comprehension, naming, fluency, repetition.

SUMMARY:
Aphasia can significantly influence a person's social relationship and quality of life. To achieve positive language outcomes, an intensive and high-repetition speech therapy is essential. However, due to the limited number of speech therapists, the intensity and frequency of training are often insufficient. Therefore, it is critical to develop other rehabilitation approaches to enhance the benefits of aphasia intervention. Virtual reality (VR) is an immersive and interactive computer simulation technology that can promote the ecological validity of speech therapy. In this study, we develop an innovative VR software for speech training to explore the effects of VR on various aspects of language outcomes.

DETAILED DESCRIPTION:
We randomly assigned study participants into 2 groups: the traditional speech therapy (ST) group and the traditional ST with additional VR training (ST+VR) group. In the ST group, each participant received 1-hour traditional ST for each session. In the ST+VR group, an additional 30-minute VR training was administered immediately after each session of traditional ST. All participants received 3 sessions of treatment every week for 3 weeks. For outcome measurement, we administered Concise Chinese Aphasia Test (CCAT) at 3 different time points: before treatment, 1 day and 3 months after the completion of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stroke with aphasia, including fluent and non-fluent types
* Age between 20~80-year-old
* Able to understand virtual reality training
* Able to cooperate with instructions and follow the rules
* Able to use the virtual reality controller and device
* Able to sign the subject's informed consent

Exclusion Criteria:

* Diagnosis of brain pathology other than stoke, such as brain tumor, Parkinson's disease, dementia
* Unable to cooperate with the instructions
* Unable to learn how to use the virtual reality controller and device
* Any medical diseases or unstable vital signs that may cause safety concern
* Severe hearing or vision impairments
* Have ever received any form of speech therapy or virtual reality training

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-04-07 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Changes Concise Chinese Aphasia Test (CCAT) scores at 1 day after treatment | Baseline and at 1 day after total treatments complete
  CCAT total scores and scores of subtests, including conversation, description, matching, listening comprehension, expression, reading recognition, sentence repetition, imitation, spontaneous writing
Changes of Concise Chinese Aphasia Test (CCAT) scores at 3 months after treatment | Baseline and at 3 months after total treatments complete
  CCAT total scores and scores of subtests, including conversation, description, matching, listening comprehension, expression, reading recognition, sentence repetition, imitation, spontaneous writing

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No